CLINICAL TRIAL: NCT01724086
Title: A Phase IIa, Open-label Trial to Evaluate the Safety, Tolerability and Efficacy of a 12 Weeks Combination Therapy of TMC647055 and TMC435 With and Without GSK23336805 With a Pharmacokinetic Enhancer With and Without Ribavirin in Chronic Genotype 1 Hepatitis C Infected Patients
Brief Title: A Study to Evaluate the Safety, Tolerability, and Effectiveness of a 12-Week Combination Therapy of TMC647055 and TMC435 With and Without GSK23336805 With a Pharmacokinetic Enhancer With and Without Ribavirin in Patients Infected With Chronic Genotype 1 Hepatitis C Virus
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR100882; TMC647055HPC2001 (Other: Janssen R&D Ireland); 2012-002555-42 (EudraCT Number)
Record Dates: First submitted 2012-09-26; First posted 2012-11-09 (Estimated); Last update posted 2016-01-11 (Estimated); Status verified 2016-01

CONDITIONS: Chronic Hepatitis C
Keywords: Chronic hepatitis C; Chronic hepatitis C-infected patients; TMC647055; TMC435; Ritonavir; Ribavirin; Genotype 1a; Genotype 1b; GSK2336805
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — 27-cyclohexyl-12,13,16,17-tetrahydro-22-methoxy-11,17-dimethyl-10,10-dioxide-2,19-methano-3,7:4,1-dimetheno-1H,11H-14,10,2,9,11,17-benzoxathiatetraazacyclo docosine-8,18(9H,15H)-dione; Simeprevir; Ritonavir; Ribavirin; peginterferon alfa-2a; GSK2336805

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (7):
- Panel 1 (Experimental): 10 chronic HCV genotype 1a (GT1a) infected treatment-naive patients/prior relapsers who will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose ritonavir and ribavirin.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: Ribavirin; Drug: Pegylated interferon alpha-2a (PegIFN)
- Panel 2 Arm 1 (Experimental): 10 chronic HCV GT1b infected treatment-naive patients/ prior relapsers will receive TMC435 + TMC647055 + low-dose ritonavir and ribavirin.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: Ribavirin; Drug: Pegylated interferon alpha-2a (PegIFN)
- Panel 2 Arm 2 (Experimental): 10 chronic HCV GT1b infected treatment-naive patients/ prior relapsers will receive TMC435 + TMC647055 + low-dose ritonavir.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: Ribavirin; Drug: Pegylated interferon alpha-2a (PegIFN)
- Panel 3 - Arm 1 (Experimental): 8 chronic HCV GT1a infected treatment naïve patients/prior relapsers will receive TMC435 + TMC647055 + low-dose ritonavir + ribavirin.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: Ribavirin; Drug: Pegylated interferon alpha-2a (PegIFN)
- Panel 3 - Arm 2 (Experimental): 8 chronically HCV GT1b infected treatment naïve patients/prior relapsers will receive TMC435 + TMC647055 + low-dose ritonavir.
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: Pegylated interferon alpha-2a (PegIFN)
- Panel 4 - Arm 1 (Experimental): 20 chronic HCV GT1a or GT1b infected treatment-naive patients/ prior relapsers will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV + GSK2336805 (30 mg once daily)
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: GSK2336805
- Panel 4 - Arm 2 (Experimental): 20 chronic HCV GT1a or GT1b infected treatment-naive patients/ prior relapsers will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV + GSK2336805 (60 mg once daily)
  Interventions: Drug: TMC647055; Drug: TMC435; Drug: Ritonavir; Drug: GSK2336805

INTERVENTIONS:
Drug: TMC647055 — Type=exact number, unit=mg, number=150, form=capsule, route=oral. 3 or 4 capsules of 150 mg will be administered once daily.
  Other Names: JNJ-42039556-AMR-G-001
Drug: TMC435 — Type=exact number, unit=mg, number=75, form=capsule, route=oral. 1 capsule of 75 mg will be administered once daily.
Drug: Ritonavir — Type=exact number, unit=mg, number=30 or 50, form=tablet or solution, route=oral. 0.375 mL or 0.625 ml (80 mg/mL) solution will be administered once daily.
Drug: Ribavirin — Type=exact number, unit=mg, number=200, form=tablet, route=oral. 5 to 6 (1000 or 1200 mg) tablets will be administered once daily, divided in 2 daily doses. Patients meeting the Follow-UP (FU) treatment criteria specified in the protocol will receive treatment 5 or 6 (depending on bodyweight) tablets of ribavirin (equivalent to 200 mg/tablet) per day, divided in 2 daily doses for an additional 12 or 36 weeks.
  Arms: Panel 1; Panel 2 Arm 1; Panel 2 Arm 2; Panel 3 - Arm 1
Drug: Pegylated interferon alpha-2a (PegIFN) — Type=exact number, unit=mcg, number=180, form=solution, route=subcutaneous injection. PegIFN 0.5 mL prefilled syringe equivalent to 180 mcg will be administered as a subcutaneous (under the skin) injection as follow-up (FU) treatment for 12 or 36 weeks based on follow-up treatment principles as described in the protocol. Patients meeting the Follow-UP (FU) treatment criteria specified in the protocol will receive treatment with Pegylated interferon alpha-2a (PegIFN) 0.5 mL prefilled syringe equivalent to 180 mcg administered as a subcutaneous (under the skin) injection for an additional 12 or 36 weeks.
  Arms: Panel 1; Panel 2 Arm 1; Panel 2 Arm 2; Panel 3 - Arm 1; Panel 3 - Arm 2
Drug: GSK2336805 — Type=exact number, unit=mg, number=30 or 60, form=tablet, route=subcutaneous injection. GSK2336805 one or two 30 mg tablet(s) taken orally (by mouth) once daily for 12 weeks.
  Arms: Panel 4 - Arm 1; Panel 4 - Arm 2

SUMMARY:
The purpose of this study is to explore the efficacy and safety of TMC647055, TMC435, and low-dose ritonavir, administered together with and without ribavirin and of TMC647055, TMC435, low-dose ritonavir administered together with GSK233680k without ribavirin in a limited number of patients with chronic hepatitis C virus (HCV) infection.

DETAILED DESCRIPTION:
This study is an open-label study (all people know the identity of the intervention) in patients who are chronically infected with hepatitis C virus (HCV) genotype-1a (GT1a) or genotype-1b (GT1b) to assess the safety, tolerability and efficacy of the coadministration of TMC647055, TMC435 and low-dose ritonavir (RTV), with and without ribavirin (RBV) and of TMC647055, TMC435, RTV administered together with GSK233680k without RBV for 12 weeks. Approximately 86 patients will be enrolled in this study. Patients enrolled in the study will be chronically infected with HCV of GT1a (n=10) or GT1b (n=20), either treatment-naive patients (ie, patients never having received PegIFN [Pegylated interferon alpha-2a at 180 mcg subcutaneous once a week], RBV, or any other approved or investigational treatment for chronic HCV infection) or patients who are relapsers to prior treatment with PegIFN /RBV (ie, "relapsers" are patients with HCV ribonucleic acid [RNA] undetectable at the last on treatment measurement of a prior PegIFN based regimen of at least 24 weeks, but HCV RNA detectable within 1 year after the last medication intake). Patients in this first part of the study will be divided over 4 panels: Panel 1 will consist of 10 chronic HCV GT1a infected treatment-naive patients/prior relapsers who will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose ritonavir and ribavirin. Panel 2 will consist of 20 chronic HCV GT1b infected treatment-naive patients/ prior relapsers who will be randomly allocated to 2 arms in a 1:1 ratio. Arm 1 (N=10) will receive TMC435 + TMC647055 + low-dose ritonavir and ribavirin. Arm 2 (N=10) will receive TMC435 + TMC647055 + low-dose ritonavir. Panel 3 will consist of 16 chronic HCV GT1a or GT1b infected treatment-naïve patients/prior relapsers who will be allocated to 2 arms: 8 HCV GT1a patients in arm 1 and 8 HCV GT1b patients in arm 2. Patients in Arm 1 will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV and RBV and patients in Arm 2 will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV. Panel 4 will consist of 40 chronic HCV GT1a or GT1b infected treatment-naïve patients/prior relapsers who will be allocated to 2 arms: each arm will consist of 20 patients of which at most 8 patients will be infected with HCV GT1b. Patients will be randomized in 1:1 ratio between the 2 arms whereby randomization will be stratified by genotype. Patients in Arm 1 will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV + GSK2336805. Patients in Arm 2 will receive 12 weeks of treatment with TMC435 + TMC647055 + low-dose RTV + GSK2336805. The planned duration of the investigational treatment is 12 weeks. Patients in Panels 1, 2, and 3 may receive follow-up treatment with 12 weeks or 36 weeks of PegIFNα + RBV; follow-up treatment principles will not apply to Panel 4 as based on available proof of concept data for such combinations, the need for an additional 12 or 36-week PegIFN/RBV follow-up therapy is expected to be very low when evaluating a 12-week regimen of 3 direct acting antiviral agents for treatment of HCV genotype 1 infections. Safety will be monitored throughout the study

ELIGIBILITY:
Inclusion Criteria:

* Documented chronic genotype 1a or genotype 1b hepatitis C virus (HCV) infection with HCV ribonucleic acid (RNA) level >100,000 IU/mL at screening
* Treatment-naive or documented prior relapser to previous treatment regimens and has stopped treatment at least 3 months before screening
* Liver biopsy within 3 years before the screening visit or elastography results available prior to first study drug dosing
* Medically stable based on physical examination, medical history, vital signs, and electrocardiogram performed at screening
* Body mass index of 18.0 to 32.0 kg/m2 and body weight more than 50 kg

Exclusion Criteria:

* Evidence of liver cirrhosis by liver biopsy or the presence of esophageal varices or a transient elastography result of >14.6 kPa within 2 years prior to first dosing
* Evidence of decompensated liver disease defined as prior history or current evidence of ascites, hepatic encephalopathy, bleeding oesophageal or gastric varices
* Evidence of any significant liver disease in addition to hepatitis C (including but not limited to hepatitis B, drug- or alcohol-related cirrhosis, autoimmune hepatitis, hemochromatosis, Wilson's disease, non-alcoholic steatohepatitis, or primary biliary cirrhosis)
* Receiving or has received any HCV-specific direct antiviral agent (HCV protease inhibitors, HCV nucleoside polymerase inhibitors, HCV non-nucleoside polymerase inhibitors, HCV NS5a inhibitors or any other HCV inhibitor targeting an HCV protein or a target involved in the HCV replication cycle
* Co-infected with human immunovirus (HIV)-1 or HIV-2, with non-genotype 1a/1b HCV, or hepatitis A or B virus infection

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2012-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with a sustained virologic response (SVR) 12 Weeks after the actual end of treatment | Week 24 (Up to 12 weeks after end-of treatment visit)
  SVR12 is defined as undetectable HCV RNA at the actual end of treatment and HCV RNA less than 25 IU/mL at 12 Weeks after the actual end of treatment.
Number of patients with adverse events | Up to Week 48 (24 weeks after end of treatment)
  Number of patients with adverse events, serious adverse events, abnormal changes in safety related laboratory values, abnormal changes in vital signs and physical examination, and abnormal echocardiogram.

SECONDARY OUTCOMES:
Number of patients with a sustained virological response (SVR at 4 and/or 24 Weeks after the actual end of treatment) | Up to 24 weeks after end of treatment
HCV RNA levels over time | Up to 24 weeks after end of treatment
Number of patients with undetectable hepatitis C virus (HCV) RNA (less than 25 IU/mL undetectable) and/or HCV RNA levels less than 25 IU/mL at all time points | Up to 24 weeks after end of treatment
Number of patients with on-treatment virologic failure | End of treatment (Week 48)
Number of patients with viral relapse | Up to 24 weeks after end of treatment
Number of patients with presence of HCV variants associated with reduced susceptibility to investigational treatment | Up to 24 weeks after end of treatment
Maximum plasma analyte concentration of TMC435 | Week 4
Minimum plasma analyte concentration of TMC435 | Week 4
Area under the plasma concentration-time curve of TMC435 | Week 4
Maximum plasma analyte concentration of TMC647055 | Week 4
Minimum plasma analyte concentration of TMC647055 | Week 4
Area under the plasma concentration-time curve of TMC647055 | Week 4
Maximum plasma analyte concentration of ritonavir (RTV) | Week 4
Minimum plasma analyte concentration of RTV | Week 4
Area under the plasma concentration-time curve of RTV | Week 4
Minimum and maximum plasma concentrations of GSK233680k | Week 4
Area under the plasma concentration-time curve of GSK233680k | Week 4

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (10):
- Belgium (7):
  - Antwerp
  - Bruges
  - Brussels
  - Edegem
  - Ghent
  - Leuven
  - Liège
- Germany (3):
  - Berlin
  - Hamburg
  - Mainz

REFERENCES:
- [Derived] Vijgen L, Thys K, Vandebosch A, Van Remoortere P, Verloes R, De Meyer S. Virology analysis in HCV genotype 1-infected patients treated with the combination of simeprevir and TMC647055/ritonavir, with and without ribavirin, and JNJ-56914845. Virol J. 2017 May 31;14(1):101. doi: 10.1186/s12985-017-0760-2. PMID 28569206